CLINICAL TRIAL: NCT02973620
Title: Expanded Access Protocol; Intermediate Size Protocol: Levosimendan Compassionate Use in Pediatric Patients With Advanced Decompensated Heart Failure Who Are Refractory to Standard Therapy
Brief Title: Levosimendan Compassionate Use in Pediatric Patients With Advanced Decompensated Heart Failure
Status: No longer available | Type: Expanded Access
Sponsor: Tenax Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TNX-LVO-02
Record Dates: First submitted 2016-11-22; First posted 2016-11-25 (Estimated); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Heart Decompensation
MeSH Terms: conditions — Heart Failure | interventions — Simendan

INTERVENTIONS:
Drug: Levosimendan — levosimendan infusion started at 0.1 mcg/kg/min for 6-12 hours, increased to 0.2 mcg/kg/min for 24-36 hours
  Other Names: Simdax

SUMMARY:
Open label study of levosimendan; planned comparison for effectiveness and safety to historic matched case controls from participating sites.

ELIGIBILITY:
General Eligibility

All patients must meet at least one of the following definitions of failed standard therapy of decompensated heart failure:

Definition for failure of standard therapy:

1. Decompensated heart failure refractory to standard therapy (Milrinone of ≥0.5mcg/kg/min for >48 hours with EF <35%) including any of the following:

   * (SaO2 - SmVO2) > 30 % or lactate >3 AND/OR
   * Need for second inotropic agent AND/OR
   * Need for positive pressure ventilation AND
   * Patient not qualifying for long term ventricular assist device support or transplant at the time of assessment.
2. Cardiogenic shock with acute decompensated heart failure (requiring positive pressure ventilation and addition of inotropic support with or without use of Milrinone with EF <35%) refractory to therapy for more than 48h including any or all of the following:

   * (SaO2 - SmVO2) > 30 % or lactate >3
   * Patient not qualifying for long term ventricular assist device support or transplant at the time of assessment.
   * Potential need for short-term mechanical circulatory support.
3. Failure to wean off ECMO support with use of standard inotropic / vasoconstrictor support.

Inclusion Criteria:

1. Male or female, ≤18 years of age with acute or acute on chronic decompensated heart failure.
2. Male or female, ≤18 years of age on ECMO support and unable to wean from ECMO support.
3. Informed Consent signed by the subject's parents or their legally acceptable representatives indicating that they understand the purpose of and procedures required for expanded access and are willing to participate in the study.
4. Patients meeting one of the following definitions of failed standard therapy of decompensated heart failure

Exclusion Criteria:

1. Patients < 36 weeks gestational age
2. Patients weighing < 2 kg
3. Obstructive cardiomyopathy, constrictive pericarditis, pericardial tamponade
4. Estimated glomerular filtration rate (eGRF) < 30 mL/min/1.73m2.
5. Known allergic reaction or sensitivity to levosimendan or excipients.
6. A history of Torsades de Pointes, uncorrectable hypo- or hyperkalemia, uncorrectable hypo- or hypercalcemia
7. Pregnant, suspected to be pregnant, or breast-feeding.
8. Inability or unwillingness of subject or legal guardian/representative to give written informed consent.

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult